CLINICAL TRIAL: NCT06690476
Title: A Open-Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of IPM514 in Patients with Esophageal Squamous Cell Carcinoma
Brief Title: Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of IPM514 in Patients with Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM514-001
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab; Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose escalation(IPM514 monotherapy) (Experimental): Drug：IPM514 Intramuscular Injection A total of 7 administrations, including 2 cycles of vaccination with each cycle at QW × 3 doses; there is a 2-weeks interval between the two cycles, then followed by a boost dose 3 weeks after the 2'nd cycle.
  Interventions: Drug: Dose escalation(IPM514 monotherapy)
- Dose expansion (IPM514 combined with tislelizumab) (Experimental): Drug：IPM514 Intramuscular Injection Drug：tislelizumab intravenous administration The usage and dosage of the tislelizumab will be based on the drug instructions. IPM514 administration is planned to be concomitant with PD-1 antibody and to be stopped after 9 doses of treatment, while the PD-1 antibody will be continuously administered for a maximum of 1 year.
  Interventions: Drug: Dose expansion (IPM514 combined with tislelizumab)
- Neoadjuvant therapy cohort(IPM514 combined with tislelizumab, cisplatin and paclitaxel) (Experimental): Drug：IPM514 Intramuscular Injection Drug：tislelizumab intravenous administration Drug：cisplatin intravenous administration Drug：paclitaxel intravenous administration In this stage, subjects will receive the treatment of IPM514 combined with Tislelizumab, cisplatin and paclitaxel. All four drugs will be administered once every 3 weeks (± 1 day). IPM514 will be administered for the first time on D0, and Tislelizumab, cisplatin and paclitaxel will be administered for the first time on D3 (the administration order: Tislelizumab - paclitaxel - cisplatin). IPM514 will be administered a total of 3 times, and PD-1 antibody, cisplatin and paclitaxel will all be administered a total of 2 times (that is, IPM514 is administered on D0/D21/D42, and Tislelizumab, paclitaxel and cisplatin are administered on D3/D24).
  Interventions: Drug: Neoadjuvant therapy cohort(IPM514 combined with tislelizumab, cisplatin and paclitaxel)

INTERVENTIONS:
Drug: Dose escalation(IPM514 monotherapy) — Drug：IPM514 Intramuscular Injection A total of 7 administrations, including 2 cycles of vaccination with each cycle at QW × 3 doses; there is a 2-weeks interval between the two cycles, then followed by a boost dose 3 weeks after the 2'nd cycle.
  Arms: Dose escalation(IPM514 monotherapy)
Drug: Dose expansion (IPM514 combined with tislelizumab) — Drug：IPM514 Intramuscular Injection Drug：tislelizumab intravenous administration The usage and dosage of the tislelizumab will be based on the drug instructions. IPM514 administration is planned to be concomitant with PD-1 antibody and to be stopped after 9 doses of treatment, while the PD-1 antibody will be continuously administered for a maximum of 1 year.
  Arms: Dose expansion (IPM514 combined with tislelizumab)
Drug: Neoadjuvant therapy cohort(IPM514 combined with tislelizumab, cisplatin and paclitaxel) — Drug：IPM514 Intramuscular Injection Drug：tislelizumab intravenous administration Drug：cisplatin intravenous administration Drug：paclitaxel intravenous administration In this stage, subjects will receive the treatment of IPM514 combined with Tislelizumab, cisplatin and paclitaxel. All four drugs will be administered once every 3 weeks (± 1 day). IPM514 will be administered for the first time on D0, and Tislelizumab, cisplatin and paclitaxel will be administered for the first time on D3 (the administration order: Tislelizumab - paclitaxel - cisplatin). IPM514 will be administered a total of 3 times, and PD-1 antibody, cisplatin and paclitaxel will all be administered a total of 2 times (that is, IPM514 is administered on D0/D21/D42, and Tislelizumab, paclitaxel and cisplatin are administered on D3/D24).
  Arms: Neoadjuvant therapy cohort(IPM514 combined with tislelizumab, cisplatin and paclitaxel)

SUMMARY:
This is a open-label, multicenter study to assess the safety, tolerability, and preliminary efficacy of IPM514 in patients with esophageal squamous cell carcinoma. This study consists of dose escalation phase (IPM514 monotherapy) ，dose expansion phase (IPM514 combined with anti-PD-1 antibody) and the neoadjuvant therapy cohort(IPM514 combined with anti-PD-1 antibody, cisplatin and paclitaxel).The dose escalation and dose expansion stages will include patients with unresectable advanced, recurrent or metastatic ESCC who have failed first-line treatment. After confirming the preliminary safety and effectiveness in the dose escalation and dose expansion stages, a neoadjuvant therapy cohort study will be developed, and resectable ESCC subjects will be included.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and agree to comply with the requirements of the study and the schedule of assessments.
2. Male or female, aged ≥ 18 years.
3. Histologically confirmed diagnosis of esophageal squamous cell carcinoma.
4. Dose escalation and dose expansion stages: After at least one line of systemic treatment (PD-1 antibody combined with platinum-based chemotherapy) has progressed or is intolerable. The following situations are regarded as the failure of the first-line standard treatment:

   * Tumor recurrence/progression during neoadjuvant/adjuvant immunotherapy combined with platinum-containing chemotherapy.
   * Patients with disease recurrence within 6 months after completing neoadjuvant/adjuvant treatment, and this neoadjuvant/adjuvant treatment is also defined as first-line treatment.
5. Dose escalation and dose expansion stages :At least one measurable lesion by RECIST v1.1, that is, the long diameter of non-lymph node lesions shown by CT or MRI is ≥10 mm or the short diameter of lymph node lesions is ≥15 mm. If the CT scan slice thickness is >5 mm, the minimum diameter of the lesion is twice the slice thickness (acceptable examination results within 28 days before signing the ICF).
6. Neoadjuvant treatment cohort: Have not received any anti-tumor treatment for esophageal cancer, including radiotherapy, chemotherapy, surgery, etc.; and plan to receive surgical treatment after the completion of neoadjuvant treatment.
7. Eastern Cooperative Oncology Group (ECOG) performance status score: 0 or 1.
8. The expected survival period is ≥12 weeks.
9. The HLA typing is HLA*A: 0201 and/or HLA*A: 1101.
10. The organ function level in the screening period must meet the following requirements (no blood transfusion or blood products, no use of hematopoietic stimulating factors and other drugs to correct the number of blood cells before the examination):

    * Absolute neutrophil count (ANC) ≥ 1.5 × 109/L;
    * Platelet count (PLT) ≥ 100 × 109/L;
    * Hemoglobin (Hb) ≥ 90 g/L;
    * Total bilirubin (TBIL) ≤ 1.5 × ULN;
    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN, ≤ 5 × ULN for those with liver metastasis;
    * Serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance rate (Cockcroft-Gault formula) ≥ 45 mL/min;
    * International normalized ratio (INR), prothrombin time (PT) ≤ 1.5 × ULN;
    * QTc interval calculated according to the Fridericia standard, ≤ 450 ms for men and ≤ 470 ms for women;
    * Urine routine/24-hour urine protein quantification: Urine protein qualitative ≤ 1+ (if urine protein qualitative ≥ 2+, then 24-hour urine protein < 1 g can be enrolled);
    * Cardiac function: Left ventricular ejection fraction ≥ 50%.
11. Eligible patients (male or female) with fertility must agree to adopt a medically approved physical contraceptive measure (such as an intrauterine device, condom, tubal or vas deferens ligation, etc.) during the trial and within 6 months after the last administration; Serum or urine HCG tests of women of childbearing age must be negative in the screening period.

Exclusion Criteria:

1. After stent implantation in esophagus; Patients who are at high risk of bleeding or perforation due to significant tumor invasion of adjacent organs (aorta or trachea).
2. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage.
3. Known allergy to the components of the study drug.
4. Prior treatment with an mRNA vaccine.
5. Subjects received major surgery within 4 weeks before the first administration or are expected to receive major surgery during the study (as judged by the investigator).
6. Dose escalation and dose expansion stages: Subjects received any anti-tumor therapy, such as chemotherapy, radiotherapy, targeted therapy, immunotherapy, and biological therapy, or any investigational therapy within 28 days or 5 half-lives (whichever is shorter but at least 14 days) of the first study drug administration:
7. Expected to use immunosuppressant drugs during the 4-week period before the first administration and during the study, except for corticosteroid nasal sprays, inhalants or systemic prednisone ≤ 10 mg/day and equivalent drugs of the same kind.
8. With a history of organ transplantation, bone marrow transplantation or hematopoietic stem cell transplantation.
9. Received live attenuated vaccines within 28 days before the first administration.
10. Dose escalation and dose expansion stages: Subjects with symptomatic, untreated or requiring continuous treatment (including corticosteroids and antiepileptic drugs) of central nervous system (CNS) metastasis (for those who have received treatment in the past, those who have been clinically stable for at least 4 weeks before enrollment, have excluded evidence of new or expanded metastasis and have discontinued steroid treatment can be enrolled; those with asymptomatic brain metastasis and do not require treatment can be enrolled.
11. 10 Dose escalation and dose expansion stages: The toxicity after previous anti-tumor treatment has not returned to the baseline or grade 0-1 as stipulated in NCI-CTCAE v5.0 (except for hair loss and pigmentation). Those with irreversible toxicities that are not expected to be aggravated by the investigational drug and can be enrolled after confirmation with the investigator.
12. With a history of autoimmune diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel diseases, etc. Type 1 diabetes mellitus, hypothyroidism that can only be controlled by replacement therapy, and skin diseases (such as vitiligo, psoriasis) that do not require systemic treatment can be enrolled.
13. With a history of immediate allergic reaction, eczema that cannot be controlled by topical corticosteroids or asthma.
14. With concomitant diseases that cannot be controlled, including but not limited to: unexplained fever > 38.5°C (subjects with tumor fever are judged by the investigator whether to include in the study), symptomatic congestive heart failure with New York Heart Association (NYHA) cardiac function classification ≥ grade 2, left ventricular ejection fraction (LVEF) < 50%, poorly controlled hypertension (systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg after treatment, and the investigator assesses that it is of clinical significance), unstable angina pectoris or acute myocardial infarction occurred within 3 months before the first administration, poorly controlled arrhythmia; patients with chronic obstructive pulmonary disease, asthma, interstitial lung disease and those with decreased pulmonary function.
15. With active infection and currently require systemic anti-infective treatment; those with active tuberculosis.
16. Known history of HIV, active Treponema pallidum infection; HBsAg positive and HBV-DNA > 500 IU/L; HCV-RNA positive.
17. Other situations judged by the investigator not suitable for participating in this study, including but not limited to having any diseases or histories that may confuse the study results or interfere with the patient's compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | up to 12 months
  Dose escalation & Dose expansion：(1) Incidence and severity of adverse events (AEs), immune-related adverse events (irAEs), serious adverse events (SAEs) assessed by NCI-CTCAE v5.0. (2) The incidence and titer of anti-drug antibodies (ADA)
The MTD, if any, and RP2D | up to 12 months
  Dose escalation & Dose expansion：IPM514 will be determined based on safety, tolerability, PK, preliminary efficacy, and other available data
PK parameter | up to 12 months
  Dose escalation & Dose expansion：mRNA quantitation in blood by qPCR
the pCR rate | up to 12 months
  Neoadjuvant Treatment Cohort：The rate of pathological complete response

SECONDARY OUTCOMES:
Objective response rate (ORR) | up to 12 months
  Dose escalation & Dose expansion：Objective response rate (ORR) per RECIST 1.1 criteria according to investigators assessment
disease control rate (DCR) | up to 12 months
  Dose escalation & Dose expansion：disease control rate (DCR) per RECIST 1.1 criteria according to investigators assessment
progression-free survival (PFS) | up to 12 months
  Dose escalation & Dose expansion：Progression free survival (PFS) rates
overall survival (OS) | up to 12 months
  Dose escalation & Dose expansion：Overall survival (OS) rates
duration of response (DOR) | up to 12 months
  Dose escalation & Dose expansion：Duration of response (DOR) per RECIST 1.1 criteria according to investigators assessment
the MPR rate | up to 12 months
  Neoadjuvant Treatment Cohort：The rate of major pathological response
the rate of R0 resection | up to 12 months
  Neoadjuvant Treatment Cohort：the rate of R0 resection
AE | up to 12 months
  Neoadjuvant Treatment Cohort：The incidence and severity of adverse events (AEs), immune-related adverse events (irAEs), and serious adverse events (SAEs) as evaluated according to NCI-CTCAE v5.0;
Surgical safety | up to 12 months
  Neoadjuvant Treatment Cohort：surgical complications within 30 days after surgery or during the postoperative hospital stay, length of hospital stay, reoperation rate, and 30-day postoperative mortality rate;
Biological responses | up to 12 months
  Neoadjuvant Treatment Cohort：(1) Lymphocyte subset analysis, including T/B/NK cell count and phenotyping of memory T cell; (2) TAA-specific T cell identification through tetramer and intracellular cytokine production via flow cytometry; (3) Immune responses of CTLs via IFN-γ ELISPOT; (4) Single-cell phenotypic analysis.
Predictive biomarkers | up to 12 months
  Neoadjuvant Treatment Cohort：including but not limited to tumor tissue antigen expression, minimal residual disease (MRD) and blood-based tumor mutational burden (bTMB)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No